CLINICAL TRIAL: NCT05502432
Title: A Prospective, Randomized, Controlled Trial for the Efficacy of Repetitive Transcranial Magnetic Stimulation in Spinocerebellar Ataxia Type 3
Brief Title: Repetitive Transcranial Magnetic Stimulation in SCA3 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., National Natural Science Foundation of China（U1505222）, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chiCTR180002013
Record Dates: First submitted 2019-09-19; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Spinocerebellar Ataxia Type 3
Keywords: Device:Active repetitive transcranial magnetic stimulation; Device:Sham repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Machado-Joseph Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Repetitive Transcranial Magnetic Stimulation(rTMS) (Active Comparator): 15 days with 1 Hz of repetitive transcranial magnetic stimulation (rTMS) with active mood.
  Interventions: Device: Active repetitive transcranial magnetic stimulation
- Sham Repetitive Transcranial Magnetic Stimulation(rTMS) (Sham Comparator): 15 days with 1 Hz of repetitive transcranial magnetic stimulation (rTMS) with sham mood.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation — Consecutive 15-day active treatment with 1 Hz of repetitive transcranial magnetic stimulation
  Arms: Active Repetitive Transcranial Magnetic Stimulation(rTMS)
Device: Sham repetitive transcranial magnetic stimulation — Consecutive 15-day sham treatment with 1 Hz of repetitive transcranial magnetic stimulation
  Arms: Sham Repetitive Transcranial Magnetic Stimulation(rTMS)

SUMMARY:
Machado-Joseph Disease (MJD) or spinocerebellar ataxia type 3 (SCA3) is the most common spinocerebellar ataxia worldwide.Repetitive transcranial magnetic stimulation (rTMS) is a form of brain stimulation therapy used to treat depression and cerebellar ataxias. In this randomized, double-blind, sham-controlled study, the investigators will evaluate whether a 15 day treatment with 1 Hz of repetitive transcranial magnetic stimulation (rTMS) can improve symptoms (motor symptoms and non-motor symptoms) in patients with MJD.

DETAILED DESCRIPTION:
Machado-Joseph Disease (MJD) or spinocerebellar ataxia type 3 (SCA3) is the most common spinocerebellar ataxia worldwide. MJD shows remarked clinical heterogeneity and presents with various clinical manifestations, including cerebellar ataxia, limb incoordination, dysarthria, sleep disorders, axonal neuropathy, dystonia, pyramidal signs and, diplopia. No effective treatment is currently available for MJD.

Repetitive transcranial magnetic stimulation (rTMS)enables non-invasive modulation of cortical excitability. rTMS targeting cerebellar structures is capable of inducing long-lasting changes in the excitability of cerebello-thalamocortical pathways.

Subjects will be randomized in two groups, one receiving a consecutive 15-day treatment with 1 Hz of repetitive transcranial magnetic stimulation and the other receiving sham stimulation with identical parameters. Patients will be clinically assessed at baseline, during intervention period at 7 days and 15 days immediate after treatment.

ELIGIBILITY:
Inclusion Criteria:

1 .Patients with detectable clinical signs and confirmed genetic diagnosis with SCA3.

2. SCA3 patients aged 20 - 80 years 3. Patients or their family members have informed consent to the study and signed relevant documents

Exclusion Criteria:

* 1. Patients who have concomitant epilepsy. 2. History of seizure or heat convulsion. 3. Patients on neuroleptics. 4. History or current unstable hypertension. 5. History of head injury or neurosurgical interventions. 6. History of any metal in the head (outside the mouth). 7. Known history of any metallic particles in the eye, implanted cardiac pacemaker, implanted neurostimulators, surgical clips (above the shoulder line) or any medical pumps.

  8. History of frequent or severe headaches. 9. History of migraine. 10. History of hearing loss. 11. History of cochlear implants 12. History of drug abuse or alcoholism. 13. Pregnancy or not using a reliable method of birth control. 14. Participation in current clinical study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
ICARS | At baseline, during intervention period at 7 days and 15 days immediate after treatment.
  The International Cooperative Ataxia Rating Scale (ICARS)

SECONDARY OUTCOMES:
BBS | At baseline, during intervention period at 7 days and 15 days immediate after treatment
  Berg Balance Scale (BBS)
SARA | At baseline, during intervention period at 7 days and 15 days immediate after treatment
  Scale for the Assessment and Rating of Ataxia (SARA)

OTHER OUTCOMES:
Tandem gait | At baseline, during intervention period at 7 days and 15 days immediate after treatment
  Tandem gait is a gait (method of walking or running) where the toes of the back foot touch the heel of the front foot at each step.
10 Metre Walk Test | At baseline, during intervention period at 7 days and 15 days immediate after treatment
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
Static Stability Test | At baseline and 15 days immediate after treatment
  Static Stability Test is a objective test use Pro-kin machine to evaluate patient's standing balance.
Pittsburgh Sleep Quality Index (PSQI) | At baseline and 15 days immediate after treatment
  The Pittsburgh Sleep Quality Index (PSQI) is the most commonly used instrument to assess the subjective sleep quality of adults in clinical and community settings
Athens Insomnia Scale (AIS) | At baseline and 15 days immediate after treatment
  The AIS is a self-reported questionnaire designed to measure the severity of insomnia based on the diagnostic criteria of the International Classification of Diseases, 10th revision (ICD-10).
Mini-Mental State Examination (MMSE) | At baseline and 15 days immediate after treatment
  In addressing cognitive screening tools, the MMSE and the MoCA are the most commonly used methods in cognitive impairment detection in both clinical and research fields.
Montreal Cognitive Assessment (MoCA） | At baseline and 15 days immediate after treatmen
  In addressing cognitive screening tools, the MMSE and the MoCA are the most commonly used methods in cognitive impairment detection in both clinical and research fields.
Hamilton Anxiety Scale (HAMA) | At baseline and 15 days immediate after treatmen
  HAMA contains 14 questions; each question includes 5 items. Responses are scored as 0 (never), 1 (mild), 2 (moderate), 3 (severe), or 4 (extremely serious). The total score of HAMA is operationally categorized as follows: no anxiety (score 0-6), mild and moderate anxiety (score 7-13), severe anxiety (score ≥ 14).
Hamilton Depression Scale (HAMD) | At baseline and 15 days immediate after treatmen
  HAMD contains 17 questions; each question includes 5 items. Responses are scored as 0 (never), 1 (mild), 2 (moderate), 3 (severe), or 4 (extremely serious). The total score of HAMD can be classified into normal (score 0-6), mild and moderate (score 7-23), severe depression (score ≥ 24).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology ,First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

REFERENCES:
- [Background] Shiga Y, Tsuda T, Itoyama Y, Shimizu H, Miyazawa KI, Jin K, Yamazaki T. Transcranial magnetic stimulation alleviates truncal ataxia in spinocerebellar degeneration. J Neurol Neurosurg Psychiatry. 2002 Jan;72(1):124-6. doi: 10.1136/jnnp.72.1.124. No abstract available. PMID 11784843
- [Background] Manor B, Greenstein PE, Davila-Perez P, Wakefield S, Zhou J, Pascual-Leone A. Repetitive Transcranial Magnetic Stimulation in Spinocerebellar Ataxia: A Pilot Randomized Controlled Trial. Front Neurol. 2019 Feb 12;10:73. doi: 10.3389/fneur.2019.00073. eCollection 2019. PMID 30809184
- [Background] Shimizu H, Tsuda T, Shiga Y, Miyazawa K, Onodera Y, Matsuzaki M, Nakashima I, Furukawa K, Aoki M, Kato H, Yamazaki T, Itoyama Y. Therapeutic efficacy of transcranial magnetic stimulation for hereditary spinocerebellar degeneration. Tohoku J Exp Med. 1999 Nov;189(3):203-11. doi: 10.1620/tjem.189.203. PMID 10674722